CLINICAL TRIAL: NCT01579500
Title: The Effect of Botulinum Toxin A in Post Spinal Cord Injury Neuropathic Pain
Brief Title: Neuropathic Pain Study With Botulinum Toxin A in Spinal Cord Injury Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of Korea Saint Paul's Hospital (Other)
Collaborators: National Health Insurance Service Ilsan Hospital (Other); Medy-Tox (Industry)
Responsible Party: Principal Investigator, Myung Eun, Chung, clinical assistant proffessor, Catholic University of Korea Saint Paul's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC12MIMV0005; 20120007154 (Other: Korea food and drug administration); suyon 2011-131 (Other: National Health Insurance Corporation Ilsan Hospital institutional review board)
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Spinal Cord Injury; Neuropathic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- botulinum toxin A (Active Comparator)
  Interventions: Drug: Botulinum toxin type A
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Botulinum toxin type A — Subcutaneous injection of botulinum toxin type A
  Arms: botulinum toxin A
Drug: normal saline — Subcutaneous injection of normal saline
  Arms: normal saline

SUMMARY:
The purpose of this study is to determine whether botulinum toxin A is effective in the treatment of neuropathic pain in spinal cord injury patients.

DETAILED DESCRIPTION:
Neuropathic pain remains a significant cause of life quality deterioration. This study includes spinal cord injury patients with refractory chronic neuropathic pain and investigates whether injection with botulinum toxin A improves pain scores.

ELIGIBILITY:
Inclusion Criteria:

* more than twenty years of age
* paraplegic or tetraplegic due to cervical and thoracic spinal cord injury
* more than 12 months since spinal cord injury and ASIA impairment scale unchanged for more than 6 months
* persistence of neuropathic pain for more than three months or remission and recurrence of neuropathic pain for more than six months
* a pain score of 40mm or more on the visual analogue scale

Exclusion Criteria:

* neuropathic pain caused by confounding factors other than spinal cord injury
* contraindicated for botulinum toxin type A
* a change in pain medication one month prior to study enrollment
* a condition involving neuromuscular junction (Ex. Eaton Lambert disease, myasthenia gravis)
* person who received botulinum toxin type A within three months prior to study enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 4 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University Saint Paul's Hospital; National Health Insurance Corporation Ilsan Hospital, Seoul, South Korea